CLINICAL TRIAL: NCT01439763
Title: Assessment of Bullying in Children With Psychiatric Symptoms: An Emergency Department Based Evaluation
Brief Title: Assessment of Bullying in Children
Acronym: ABC
Status: Completed | Type: Observational
Sponsor: New York City Health and Hospitals Corporation (Other)
Responsible Party: Principal Investigator, Muhammad Waseem, Research Director, Emergency Medicine, New York City Health and Hospitals Corporation
Other Study IDs: 10-027
Record Dates: First submitted 2011-09-21; First posted 2011-09-23 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Problematic Behavior in Children
Keywords: Bullies; Bully victims; Psychiatric symptoms
MeSH Terms: conditions — Bullying

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The specific aims of this study are:

* To determine the prevalence of bullying in children who present to the ED with behavioral symptoms
* To assess mental health diagnoses and their relationship to type, severity and frequency of bullying behaviors, as well as demographic and psychosocial correlates (socioeconomic status, stress and support) and their relationship to type, severity and frequency of bullying (bullies versus victims).
* To explore the attitudes, values, triggering events and potential solutions using qualitative methods
* To gain greater insight into the patient experience and perceptions of the bullying events

DETAILED DESCRIPTION:
This is a mix method study which has both qualitative and quantitative components.

* Data Collection sheet
* Qualitative Measurement
* Quantitative Measurement
* Data Collection sheet

  1. Demographic information (Date of birth, gender, race/ethnicity)
  2. Assessment of socioeconomic status (Type of Insurance, Zip Code, Parent education level, Parent type of work)
  3. Child physical attributes (Appearance, Weight, Height, Percentiles & BMI, Assisted Devices, Disabilities)
  4. Academic performance (Whether grades are age appropriate, previous grade results
  5. Extra-curricular activities (Questions include do you participate in sports? Are you member of any sport team? Are you member of any club?)

Qualitative Measurement

In order to understand bullying and victimization, a brief qualitative interview will be conducted by the principal investigator and his team. These questions may provide insights into the dynamics of bullying.

Quantitative Measurement

Following measurement scales will be used in the assessment of children with bullying Bullying → Olweus Bullying Questionnaire Child behavior → Achenbach Child Behavior Checklist Stress, life events and adversities → Adolescent Perceived Events Scale (APES) Social support → Child and Adolescent Social Support Scale (Malecki 2000) Social status → MacArthur Scale of Subjective Social Status Family Structure → A documentation of family structure and dynamics Mental health status → Psychiatric evaluation

ELIGIBILITY:
Inclusion Criteria:

* Children with psychiatric or behavioral problem(s) age 8-18 years referred from the school to the ED
* Parents willing to provide informed consent and child providing assent

Exclusion Criteria:

* Actively violent behavior
* Child abuse
* Parents or children refuse to participate

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children 8-18 years of age referred from school to the Emergency Department due to Behavior Problems
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2011-09 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Bullying | last one year
  Bullying incidents

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Waseem, MD, Principal Investigator — Lincoln Medical & Mental Health Center, Bronx New York
Locations (1):
- Lincoln Medical & Mental Health Center, The Bronx, New York, United States

REFERENCES:
- [Background] Nansel TR, Overpeck M, Pilla RS, Ruan WJ, Simons-Morton B, Scheidt P. Bullying behaviors among US youth: prevalence and association with psychosocial adjustment. JAMA. 2001 Apr 25;285(16):2094-100. doi: 10.1001/jama.285.16.2094. PMID 11311098
- [Background] Analitis F, Velderman MK, Ravens-Sieberer U, Detmar S, Erhart M, Herdman M, Berra S, Alonso J, Rajmil L; European Kidscreen Group. Being bullied: associated factors in children and adolescents 8 to 18 years old in 11 European countries. Pediatrics. 2009 Feb;123(2):569-77. doi: 10.1542/peds.2008-0323. PMID 19171624
- [Background] Olweus D. Bullying at school: basic facts and effects of a school based intervention program. J Child Psychol Psychiatry. 1994 Oct;35(7):1171-90. doi: 10.1111/j.1469-7610.1994.tb01229.x. No abstract available. PMID 7806605
- [Background] Nansel TR, Craig W, Overpeck MD, Saluja G, Ruan WJ; Health Behaviour in School-aged Children Bullying Analyses Working Group. Cross-national consistency in the relationship between bullying behaviors and psychosocial adjustment. Arch Pediatr Adolesc Med. 2004 Aug;158(8):730-6. doi: 10.1001/archpedi.158.8.730. PMID 15289243
- [Background] Luukkonen AH, Rasanen P, Hakko H, Riala K; STUDY-70 Workgroup. Bullying behavior in relation to psychiatric disorders and physical health among adolescents: a clinical cohort of 508 underage inpatient adolescents in Northern Finland. Psychiatry Res. 2010 Jun 30;178(1):166-70. doi: 10.1016/j.psychres.2010.04.022. Epub 2010 May 14. PMID 20471097
- [Background] Sourander A, Ronning J, Brunstein-Klomek A, Gyllenberg D, Kumpulainen K, Niemela S, Helenius H, Sillanmaki L, Ristkari T, Tamminen T, Moilanen I, Piha J, Almqvist F. Childhood bullying behavior and later psychiatric hospital and psychopharmacologic treatment: findings from the Finnish 1981 birth cohort study. Arch Gen Psychiatry. 2009 Sep;66(9):1005-12. doi: 10.1001/archgenpsychiatry.2009.122. PMID 19736357
- [Background] Wolke D, Woods S, Bloomfield L, Karstadt L. Bullying involvement in primary school and common health problems. Arch Dis Child. 2001 Sep;85(3):197-201. doi: 10.1136/adc.85.3.197. PMID 11517098
- [Background] Jansen DE, Veenstra R, Ormel J, Verhulst FC, Reijneveld SA. Early risk factors for being a bully, victim, or bully/victim in late elementary and early secondary education. The longitudinal TRAILS study. BMC Public Health. 2011 Jun 6;11:440. doi: 10.1186/1471-2458-11-440. PMID 21645403
- [Background] Due P, Damsgaard MT, Lund R, Holstein BE. Is bullying equally harmful for rich and poor children?: a study of bullying and depression from age 15 to 27. Eur J Public Health. 2009 Oct;19(5):464-9. doi: 10.1093/eurpub/ckp099. Epub 2009 Jul 8. PMID 19587227
- [Background] Due P, Merlo J, Harel-Fisch Y, Damsgaard MT, Holstein BE, Hetland J, Currie C, Gabhainn SN, de Matos MG, Lynch J. Socioeconomic inequality in exposure to bullying during adolescence: a comparative, cross-sectional, multilevel study in 35 countries. Am J Public Health. 2009 May;99(5):907-14. doi: 10.2105/AJPH.2008.139303. Epub 2009 Mar 19. PMID 19299676
- [Background] Compas BE, Davis GE, Forsythe CJ, Wagner BM. Assessment of major and daily stressful events during adolescence: the Adolescent Perceived Events Scale. J Consult Clin Psychol. 1987 Aug;55(4):534-541. doi: 10.1037/0022-006X.55.4.534. No abstract available. PMID 3624609
- [Derived] Waseem M, Boutin-Foster C, Robbins L, Gonzalez R, Vargas S, Peterson JC. Perspectives on bullying among children who present to the emergency department with behavioral misconduct: a qualitative study. Pediatr Emerg Care. 2014 Nov;30(11):793-7. doi: 10.1097/PEC.0000000000000261. PMID 25343737